CLINICAL TRIAL: NCT00595881
Title: Emergency Bedside Ultrasound for the Evaluation of Soft Tissue Infections in the Pediatric Emergency Department
Brief Title: Emergency Bedside Ultrasound for Pediatric Soft Tissue Infections
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Other Study IDs: 2007-6-5388
Record Dates: First submitted 2008-01-07; First posted 2008-01-16 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2012-12-31 (Estimated); Status verified 2012-02

CONDITIONS: Abscess
Keywords: Bedside emergency ultrasound; Abscess; Cellulitis; Soft tissue infection; Methicillin resistant staphylococcus aureus (MRSA)
MeSH Terms: conditions — Abscess; Cellulitis; Soft Tissue Infections

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ultrasound: One group of patients will undergo emergency bedside ultrasound in addition to the clinical examination.
  Interventions: Device: Bedside emergency ultrasound

INTERVENTIONS:
Device: Bedside emergency ultrasound — Ultrasound will be performed on the lesion in question.

SUMMARY:
The purpose of this study is to determine if soft tissue infections in pediatric patients can be more accurately diagnosed (i.e. the presence of a drainable abscess) with the addition of bedside ultrasound to the clinical examination compared to the clinical examination alone.

DETAILED DESCRIPTION:
Skin and soft tissue infections, particularly abscesses caused by community-acquired methicillin resistant Staphylococcus aureus (CA-MRSA) are a growing public health problem. The treatment of a skin abscess usually requires incision and drainage or needle aspiration. In addition to providing definitive therapy, appropriate drainage can allow for organism identification and antibiotic susceptibility testing should antibiotics be utilized. A skin cellulitis, which is treated with systemic antibiotics and supportive care alone, may be hard to distinguish from an abscess, as both have similar clinical features. Therefore, as the presence or absence of purulent material may be difficult to determine, children may undergo an unnecessary drainage procedure. If drainage is avoided, the patient may require a subsequent ED visit if the diagnosis is missed on initial examination. This can lead to worsened clinical outcome, an extra financial burden for the family, and added emotional distress for the patient.

Bedside emergency ultrasound (EUS), which has been used since the mid-1980s is being used in adults to detect fluid collections such as soft tissue abscesses. Studies in adult patients have shown that EUS adds useful information to the history and physical examination and may even alter physicians' clinical impressions and management of patients. Currently, it is not known whether children represent a different population for EUS than adults and how EUS would perform in the pediatric outpatient setting. With improved diagnosis of soft tissue infections, better epidemiologic data about organism prevalence, improved and more prompt treatment, and more appropriate use of antibiotic therapy can be done.

To date, no study exists evaluating its utility specifically for the evaluation of soft tissue infections in pediatric patients. The goal of this study is to evaluate the test characteristics of EUS in pediatric patients presenting with evidence of soft tissue infection.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of at least one of the following: skin elevation, induration, tenderness, fluctuance, or history of purulent drainage from the lesion

Exclusion Criteria:

* Suspected paronychia or felon
* Lesion involving the face, perirectal, or vaginal area
* Surgical wound infection
* Underlying immunodeficiency
* Non-soft tissue infectious mass (e.g. lymphadenitis)
* Suspected non-infectious mass (e.g. hernia, lymph node)

Ages: 2 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients will be recruited from the emergency department at a tertiary care children's hospital with annual census of 78,000 patients per year.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Actual)
Dates: Start 2008-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Alpern, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Marin JR, Dean AJ, Bilker WB, Panebianco NL, Brown NJ, Alpern ER. Emergency ultrasound-assisted examination of skin and soft tissue infections in the pediatric emergency department. Acad Emerg Med. 2013 Jun;20(6):545-53. doi: 10.1111/acem.12148. PMID 23758300

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited over a 22 month period
Period: Overall Study
Arm/Group | Ultrasound
Started | 420
Completed | 420
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ultrasound
Number analyzed (Participants) | 420
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 420
  Between 18 and 65 years | 0
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 7.8 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218
  Male | 202
Region of Enrollment [Number; unit: participants]
  United States | 420

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity and Specificity of Bedside Emergency Ultrasound When Added to the Clinical Examination Compared With Clinical Examination Alone.
Description: The sensitivity and specificity of clinical examination with the addition of bedside emergency ultrasound will be compared against that of clinical examination alone.The number of lesions determined to actually have a drainable fluid collection will serve as the denominator in the calculation of sensitivity, and the number of lesions correctly identified as having a drainable fluid collection by clinical exam plus ultrasound and clinical exam alone, respectively, will serve as the numerator.The number of lesions determined to not have a drainable fluid collection will serve as the denominator in the calculation of specificity, and the number of lesions correctly identified as not having a drainable fluid collection by clinical exam plus ultrasound and clinical exam alone, respectively, will serve as the numerator. Significance will be defined as a 95% confidence interval surrounding the differences between the two groups for sensitivity and specificity that does not include 0.
Time Frame: 18 mos
Population: Assuming a baseline sensitivity of clinical exam alone similar to that previously published (86%), type 1 error rate 0.05, and intraclass correlation coefficient of 0.5 for lesions within patients, we estimated a sample size of 393 lesions would provide 80% power to detect at least a 9% difference in the sensitivity of CE+EUS compared to CE alone.
Measure: Number (95% Confidence Interval); unit: Ratio as a percentage
Groups:
- Clinical Exam Alone: Patients will have data collected from their clinical examination alone
- Clinical Exam+ Ultrasound: Patients will have data collected following the addition of a bedside ultrasound performed to the clinical exam.
Arm/Group | Clinical Exam Alone | Clinical Exam+ Ultrasound
Number analyzed (Participants) | 420 | 420
Ratio as a percentage
  Sensitivity | 94.7 [90.2 to 97.9] | 93.1 [88.6 to 97.0]
  Specificity | 84.2 [74.7 to 91.7] | 81.4 [70.8 to 90.3]
Statistical Analysis 1: Comparison: Clinical Exam Alone vs Clinical Exam+ Ultrasound; See sample size calculations already entered. Null hypothesis is that there is no difference in the sensitivity or specificity of clinical exam alone compared with clinical exam+ultrasound; Test type: Superiority or Other; Mixed effects logistic regression — We calculated the differences between the sensitivities and specificities. The difference in sensitivity between the clinical exam alone vs clinical exam + ultrasound was -1.7% (-3.4%, 0%). The difference in specificity was -2.8% (-9.7%, 4.1%); We used the bootstrap method to obtain valid confidence intervals and compare sensitivity and specificity for the 2 tests; Difference in sensitivity = -1.7, 95% CI 2-sided [-3.4 to 0] — The clinical exam alone was compared to the clinical exam + ultrasound
Statistical Analysis 2: Comparison: Clinical Exam Alone vs Clinical Exam+ Ultrasound; as previously described for sensitivity; Test type: Superiority or Other; Statistical significance was defined as a CI surrounding the difference between groups not including 0; as previously described for sensitivity; Difference in specificity = -2.8, 95% CI [-9.7 to 4.1]

ADVERSE EVENTS:
Arm/Group | Ultrasound
Serious Adverse Events (participants affected / at risk) | 0/420
Other Adverse Events (participants affected / at risk) | 0/420

LIMITATIONS AND CAVEATS:
Potential misclassification of lesions based on reference standard. Biased lesion outcome, as ultrasound results were not incorporated into patient care.

Single institution

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes